CLINICAL TRIAL: NCT05060224
Title: Low-Level Laser Therapy: an Efficient Supplement to Treatments of Vulvar Lichen Sclerosus to Improve Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kolding Sygehus (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18/27286
Record Dates: First submitted 2021-09-16; First posted 2021-09-29 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-09

CONDITIONS: Quality of Life

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Low Level Laser (Experimental): EasyLaser: Low Level Laser 808 nm and 500 mW. The first four treatments where planned as two treatments per week. The remaining six treatments where planned as once a week.
  Interventions: Device: EasyLaser: Low Level Laser therapy

INTERVENTIONS:
Device: EasyLaser: Low Level Laser therapy

SUMMARY:
Objectives: The aim of this study was to investigate whether Low Level Laser therapy (LLLT) can improve the quality of life in women with Lichen Sclerosus (LS) and insufficient topical treatment.

Methods: In a clinical trial study conducted between January 2016 and July 2018, the investigators included 100 women with LS with insufficient topical treatment. All participants received ten LLLT treatments (808 nm and 500 mW) over a period of 8 weeks. The first four treatments where planned as two treatments per week. The remaining six treatments where planned as once a week. The effect was monitored by a Danish health-related quality of life tool (HRQoL test).

DETAILED DESCRIPTION:
Hundred participants with LS were included in a clinical trial at Lillebaelt Hospital, Denmark in the period from 02.01.2016 to 08.01.2018. The participants were informed about the purpose of research and the fact that LLLT was not standard-of-care treatment in our out-patient clinic. All participants who declined to take part in the study received standard-of-care treatment (topical steroid or topical calcineurin inhibitors) according to Danish national guidelines. Participants enrolled in the study received both standard-of-care treatment and LLLT.

The participants received 10 LLLT treatments of 808 nm and 500mW. Every treatment was with a duration of 10 minutes. The first four treatments where planned as two treatments per week. The remaining six treatments where planned as once a week due to logistic considerations. The participants received the LLLT treatment while lying in the same position as during a gynecological examination. The light waves were placed 10 centimeters from the anogenital area covering the symptomatic area. If the participants had symptoms from both the vulva and the area around the rectum, the light were replaced after 10 minutes of treatment making sure no area were treated twice. All patients were recommended to continue their topical treatment during the study period. A Danish health-related quality of life tool (DoloTest®) was used to evaluate the effect of the treatment. The HRQoL test is a validated Danish tool developed for pain patients. It is validated against the Medical Outcomes Study Short Form Surveys (SF36TM). The HRQoL test requires little time and is therefore easy to use in a clinical setting. It is composed of eight domains arranged in a radar plot; pain, problems sleeping, reduced social life, low spirit, reduced energy and physical strength, problems at work, problems with more strenuous physical activity, and problems with light physical activity. Starting with the domain pain the patient marks every domain horizontally moving clockwise and thereby creates a graphic illustration, which helps the physician and the participant to understand the impact of the condition. The larger the shaded area the more the patient feels affected. Every mark represents a score. The maximum score of the HRQoL test is the total sum of the eight domains multiplied by 100, the maximum score being 800. The participants completed the HRQoL test before first LLLT treatment and after the last treatment. A written informed consents was obtained from all patients enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with lichen sclerosus either clinically or by histopathological verification
* Age ≥ 18 years
* No significant relief in symptoms despite of topical treatment with potent steroids or calcineurin inhibitors

Exclusion Criteria:

* Age < 18 years
* History of vulvar intraepithelial neoplasi

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Quality of life, scale | up to 10 weeks
  Danish health-related quality of life tool

CONTACTS AND LOCATIONS:
Overall Officials: Annemette Lykkebo, MD, Study Chair — Sygehus Lillebælt, Kolding.

IPD SHARING:
Plan to Share IPD: No
Not planned.